CLINICAL TRIAL: NCT01292798
Title: Open Label, Phase I/II, Residual Edema Evaluation With 0.5mg and 2.0mg Ranibizumab Formulations (REEF)
Brief Title: Ranibizumab 0.5mg and 2.0mg to Treat Diabetic Macular Edema in Patients With Poor Response to Bevacizumab
Acronym: REEF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: California Retina Consultants (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FVF4978s
Record Dates: First submitted 2011-02-07; First posted 2011-02-10 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetes; Macula; Edema; Retina
MeSH Terms: conditions — Diabetes Mellitus; Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5mg and 2.0mgRanibizumab (Experimental): Three consecutive intravitreal ranibizumab 0.5mg injections followed by three consecutive intravitreal ranibizumab 2.0mg injections if specific criteria is met.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.05ml of 0.5mg or 2.0mg ranibizumab injected intravitreally
  Other Names: Lucentis

SUMMARY:
This is an open-label, Phase I/II study of intravitreally administered ranibizumab either 0.5-mg and/or 2.0-mg in subjects with clinical, angiographic, and ocular coherence tomography (OCT) evidence of diabetic retinopathy with associated diabetic macular edema following bevacizumab therapy. Thirty patients will be enrolled in this study.

Consented, enrolled subjects will receive multiple open-label intravitreal injections of 0.5 mg ranibizumab administered every 30 days (±7 days) for 3 injections during the mandatory treatment phase (Day 0, Month 1, and Month 2).

Subjects with complete resolution of diabetic macular edema after 3 intravitreal injections of 0.5 mg ranibizumab will be treated as necessary with 0.5 mg ranibizumab to treat recurrent macular edema for an additional 9 months (12 months from Day 0). The intent is to administer additional ranibizumab treatment if there is evidence of disease activity documented on OCT (e.g., intra-retinal fluid, subretinal fluid and/or cystic changes).

Subjects with residual diabetic macular edema following 3 intravitreal injections of 0.5 mg ranibizumab will be receive 3 intravitreal injections of 2.0 mg ranibizumab administered every 30 days (±7 days) for 3 injections at the Month 3, Month 4, and Month 5 study visits.

Beginning at the Month 6 study visit, subjects with complete resolution of diabetic macular edema following 3 intravitreal injections of 2.0 mg ranibizumab will treated as necessary with 2.0 mg ranibizumab injections only to treat recurrent macular edema for an additional 6 months (12 months from Day 0).

Subjects with residual diabetic macular edema following 3 consecutive intravitreal injections of 2.0 mg ranibizumab will be treated as necessary with 2.0 mg ranibizumab to treat persistent or recurrent macular edema for an additional 6 months (12 months from Day 0). Focal photocoagulation or intravitreal triamcinolone may be administered at the physician's discretion as an adjunct to ranibizumab injections beginning at Month 6 through Month 12 of the study.

All subjects will make monthly visits for 12 months for evaluation of safety and efficacy. All subjects will have their first injection of ranibizumab on Day 0 and undergo a safety visit one week (±2 days) after the first injection. At subsequent visits, the subject will have a safety evaluation at the monthly scheduled follow-up visit prior to any intravitreal injection. Subjects will be contacted by the site personnel 1-2 days after each injection to elicit reports of decreased vision or pain or unusual new ocular symptoms in the study eye.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Diagnosis of diabetes mellitus (type 1 or 2)Any one of the following will be considered to be sufficient evidence that diabetes is present:Current regular use of insulin for treatment of diabetes or current regular use of oral anti-hyperglycemia agent for the treatment of diabetes
* Clinical evidence of retinal thickening due to macular edema involving the center of the macula, associated with diabetic retinopathy.
* Previous history of two consecutive intravitreal bevacizumab injections for the treatment of diabetic macular edema with documented incomplete resolution of central subfield thickening by OCT (consecutive injections administered < 7 weeks apart and within the past 12 months).
* Central diabetic macular edema present on clinical examination and OCT testing with central 1mm subfield thickness greater than 300 microns as measured on SD-OCT.
* Visual acuity score greater than or equal to 19 letters (20/400) and less than or equal to 73 letters (20/40) by the ETDRS visual acuity protocol.
* Media clarity, pupillary dilation and patient cooperation sufficient to allow OCT testing and retinal photography

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or known to be pregnant; also pre-menopausal women not using adequate contraception.
* Participation in another ocular investigation or trial simultaneously
* Blood pressure > 180/110 (systolic above 180 OR diastolic above 110)
* Any condition that, in the opinion of the investigator, would preclude participation in the study (e.g. chronic alcoholism, drug abuse)
* Evidence of vitreoretinal interface abnormality after ocular exam or OCT that may be contributing to the macular edema
* An eye that, in the investigator's opinion, has no chance of improving in visual acuity following resolution of macular edema (e.g. presence of subretinal fibrosis or geographic atrophy)
* Presence of another ocular condition that may affect the visual acuity or macular edema during the course of the study (e.g. AMD, uveitis, Irvine-Gas)
* Evidence of neovascularization of the iris or retina
* Evidence of central atrophy or fibrosis in the study eye
* Presence of substantial cataract, one that might decrease the vision by 3 or more lines of vision at sometime during the study.
* History of vitreous surgery in the study eye
* History of cataract surgery within 6 months of enrollment.
* History of YAG capsulotomy within 2 months of enrollment.
* Visual acuity <20/400 in the fellow eye
* Uncontrolled glaucoma (pressure >30) despite treatment with glaucoma medications.
* History of cerebral vascular accident or myocardial infarction within 3 months prior to Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dante Pieramici, MD, Principal Investigator — California Retina Consultants
Locations (5):
- United States (5):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Oxnard, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - Retina Institute of Hawai'i, Honolulu, Hawaii

REFERENCES:
- [Derived] Dhoot DS, Pieramici DJ, Nasir M, Castellarin AA, Couvillion S, See RF, Steinle N, Bennett M, Rabena M, Avery RL. Residual edema evaluation with ranibizumab 0.5 mg and 2.0 mg formulations for diabetic macular edema (REEF study). Eye (Lond). 2015 Apr;29(4):534-41. doi: 10.1038/eye.2014.338. Epub 2015 Jan 30. PMID 25633882

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.0 mg Ranibizumab: Subjects who presented with persistent DME at month 3 following 3 months of monthly 0.5 mg ranibizumab injections received 3 monthly injections of 2.0 mg Ranibizumab.
Period: Overall Study
Arm/Group | 2.0 mg Ranibizumab
Started | 43
Persistent DME After 3 Months | 29 (Subjects with persistent DME after 3 monthly injections of 0.5 mg of ranibizumab)
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 2.0 mg Ranibizumab
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change in Visual Acuity Scores at Month 6 Compared to Baseline
Description: To determine the mean change in the best-corrected visual acuity on an ETDRS visual acuity chart at a starting distance of 4 meters from baseline to 6 months.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 0.5mg and 2.0mgRanibizumab
Number analyzed (Participants) | 43
letters
  Baseline | 58.8 (9.7)
  6 months | 67.6 (9.3)
  Change from Baseline to 6 months | 8.8 (9.3)

2. Secondary Outcome: Mean Change in 1-mm Central Subfield (CST) Thickness as Measured by OCT at Month 6 Compared to Baseline
Description: To determine the mean change in central 1-mm subfield thickness as measured by spectral-domain OCT from baseline to 6 months .
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | 0.5mg and 2.0mgRanibizumab
Number analyzed (Participants) | 43
microns
  Baseline | 500.6 (129.1)
  6 months | 335.2 (91.5)
  Change from Baseline to 6 months | -165.4 (91.5)

3. Secondary Outcome: Qualitative Assessment of Diabetic Macular Edema (DME)
Description: To compare the percentage of subjects with compete or partial/no resolution of diabetic macular edema in response to the ranibizumab 0.5 and 2.0 mg doses.
Time Frame: Baeline and 6 months
Population: At 6 months, 18 out of the 43 subjects (42%) showed complete resolution of DME. 25 out of the 43 subjects (58%) showed partial or no resolution of DME at 6 months.
Measure: Number; unit: percentage of participants
Arm/Group | 0.5mg and 2.0mgRanibizumab
Number analyzed (Participants) | 43
percentage of participants
  complete resolution | 42
  partial/no resolution | 58

ADVERSE EVENTS:
Arm/Group | 2.0 mg Ranibizumab
Serious Adverse Events (participants affected / at risk) | 1/43
Other Adverse Events (participants affected / at risk) | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.0 mg Ranibizumab (N=43)
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes